CLINICAL TRIAL: NCT01140295
Title: Polyethylene Glycol Powder Solution vs Senna for Bowel Preparation for Colonoscopy in Children: A Prospective, Randomized, Investigator-Blinded Trial.
Brief Title: Bowel Preparation for Colonoscopy in Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Petar Mamula, Director, Endoscopy, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2006-10-5004
Record Dates: First submitted 2010-06-01; First posted 2010-06-09 (Estimated); Results first posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Colonoscopy Preparation
Keywords: Preparation; Pediatric; Colonoscopy
MeSH Terms: interventions — Polyethylene Glycols; Sennosides; polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1, Miralax (Active Comparator): Miralax colonoscopy preparation
  Interventions: Drug: polyethylene glycol, senna
- 2, senna (Active Comparator): Senna colonoscopy preparation
  Interventions: Drug: polyethylene glycol, senna

INTERVENTIONS:
Drug: polyethylene glycol, senna — Senna dosage: Age 6-12 years: 3 teaspoons or 3 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. Age >12 years: 6 teaspoons or 6 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. A Fleet's rectal enema is administered on the morning of the procedure.
  Miralax at a dose of 1.5 grams/kg divided twice a day for two days; maximum of 51 grams per dose. Dissolve each 17 grams (1 capful) PEG-P in 240 mL water or other beverage according to the manufacturer's direction and to give the appropriate amount of PEG solution twice a day for two days.
  Other Names: Miralax; Senna

SUMMARY:
The primary objective of this study is to determine whether Miralax results in a more efficacious preparation as compared to senna for pediatric colonoscopy.

DETAILED DESCRIPTION:
Study subjects will be randomized in two groups: Group one will receive 1.5 g/kg of Miralax orally the day before procedure and one day of clear liquid diet, while subjects in Group 2 will receive two doses of senna the day before procedure with two days of liquid diet (one day full liquid and one day clear liquid diet). On the day of the procedure parents/subjects will complete a questionnaire regarding prep compliance and adverse events. Electrolytes will be obtained prior to colonoscopy to monitor for electrolyte imbalance. Endoscopists will assess preparation for colonoscopy using validated cleanliness scale (Aronchick scale).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age 6-21 yrs for senna, PEG-P groups
2. Subjects age 13-21 yrs for NaP group
3. First time colonoscopy
4. Patient weight <70 kg for PEG-P group (to not exceed 51 grams/dose)

Exclusion Criteria:

1. Chronic renal, liver, or heart failure
2. Chronic constipation
3. Patients on the GI inpatient or consult service.
4. Subjects taking senna or PEG on a regular basis for laxative reasons.
5. Pregnant or lactating females

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Petar Mamula, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Terry NA, Chen-Lim ML, Ely E, Jatla M, Ciavardone D, Esch S, Farace L, Jannelli F, Puma A, Carlow D, Mamula P. Polyethylene glycol powder solution versus senna for bowel preparation for colonoscopy in children. J Pediatr Gastroenterol Nutr. 2013 Feb;56(2):215-9. doi: 10.1097/MPG.0b013e3182633d0a. PMID 22699838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at The Children's Hospital of Philadelphia Main site Endoscopy suite from September 2010 to April 2011.
Pre-assignment Details: 365 patients were screened. 98 were eligible according to inclusion/exclusion criteria. 41 declined participation. criteria. Of the 57 eligible patients 33 were enrolled when the study was prematurely terminated.
Groups:
- 1, Miralax: Miralax colonoscopy preparation
  Miralax (PEG-P) at a dose of 1.5 grams/kg divided twice a day for two days; maximum of 51 grams per dose. Dissolve each 17 grams (1 capful) PEG-P in 240 mL water or other beverage according to the manufacturer's direction and to give the appropriate amount of PEG solution twice a day for two days.
- 2, Senna: Senna colonoscopy preparation
  polyethylene glycol, senna : Senna dosage: Age 6-12 years: 3 teaspoons or 3 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. Age >12 years: 6 teaspoons or 6 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. A Fleet's rectal enema is administered on the morning of the procedure.
Period: Overall Study
Arm/Group | 1, Miralax | 2, Senna
Started | 17 | 16
Completed | 16 | 14
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- 1, Miralax: Miralax colonoscopy preparation
  polyethylene glycol, senna : Senna dosage: Age 6-12 years: 3 teaspoons or 3 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. Age >12 years: 6 teaspoons or 6 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. A Fleet's rectal enema is administered on the morning of the procedure.
  Miralax at a dose of 1.5 grams/kg divided twice a day for two days; maximum of 51 grams per dose. Dissolve each 17 grams (1 capful) PEG-P in 240 mL water or other beverage according to the manufacturer's direction and to give the appropriate amount of PEG solution twice a day for two days.
- 2, Senna: Senna colonoscopy preparation
  polyethylene glycol, senna : Senna dosage: Age 6-12 years: 3 teaspoons or 3 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. Age >12 years: 6 teaspoons or 6 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. A Fleet's rectal enema is administered on the morning of the procedure.
  Miralax at a dose of 1.5 grams/kg divided twice a day for two days; maximum of 51 grams per dose. Dissolve each 17 grams (1 capful) PEG-P in 240 mL water or other beverage according to the manufacturer's direction and to give the appropriate amount of PEG solution twice a day for two days.
- Total: Total of all reporting groups
Arm/Group | 1, Miralax | 2, Senna | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 16 | 33
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 12 (1.3) | 15 (1.2) | 14.5 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Colon Preparation
Description: Percentage of patients with excellent or good colonoscopy preparation. The efficacy of preparation is measured by using a validated colon cleanliness scale which has 5 different levels (Aronchik scale). Levels 1 and 2, which encompass excellent and good colonoscopy preparation, are routinely recognized as adequate preparation allowing for successful completion of colonoscopy. Levels 3-5 describe incomplete or poor preparation. These levels are associated with significant residual stool encountered at the time of colonoscopy.
Time Frame: The outcome measure will be assessed once one day after the completion of colonoscopy preparation
Measure: Number; unit: percentage of patients
Arm/Group | 1, Miralax | 2, Senna
Number analyzed (Participants) | 17 | 16
percentage of patients | 88 | 28

2. Secondary Outcome: Proportion of Patients With Abnormal Electrolyte Levels
Description: The outcome measure was comparison of the proportions of patients who had abnormal electrolyte levels between two groups of patients, Miralax and senna.
  Sodium, potassium, chloride, and carbon dioxide levels were measured in mmol/L while urea nitrogen, creatinine, glucose, calcium, magnesium, and phosphorus were measured in mg/dL. Each of these values has a reference range which varies with patients' age and sex. Minimal change of one point above or below normal reference range was dismissed as clinically insignificant. Abnormal creatinine levels were rechecked through glomerular filtration rate calculation to determine if there was any compromise in renal function since abnormal creatinine level does not mean there is renal dysfunction nor that the level is clinically significant.
Time Frame: The outcome measure will be assessed once one day after the completion of colonoscopy preparation
Measure: Number; unit: Proportion of patients
Groups:
- 2, Senna: Senna colonoscopy preparation
  Senna dosage: Age 6-12 years: 3 teaspoons or 3 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. Age >12 years: 6 teaspoons or 6 tablets by mouth 2 nights before endoscopy and 1 night before endoscopy. A Fleet's rectal enema is administered on the morning of the procedure.
Arm/Group | 1, Miralax | 2, Senna
Number analyzed (Participants) | 17 | 16
Proportion of patients | 0 | 0

ADVERSE EVENTS:
Arm/Group | 1, Miralax | 2, Senna
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

LIMITATIONS AND CAVEATS:
Early termination due to poor efficacy in one of the study arms (senna preparation).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No